CLINICAL TRIAL: NCT02197793
Title: Activating Treatment as Prevention Through Community Mobilization in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Witwatersrand, South Africa (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-13575
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Mobilization Program (Experimental): Intervention activities will map onto six mobilization domains identified as key components for communities to mobilize for change around testing, linkage and retention in care (Treatment as Prevention (TasP)).
  Interventions: Behavioral: Community Mobilization Program
- Control Arm (No Intervention): The control arm does not receive the Community Mobilization Intervention.

INTERVENTIONS:
Behavioral: Community Mobilization Program
  Arms: Community Mobilization Program

SUMMARY:
The purpose of this study is to evaluate the impact of a community mobilization intervention on the uptake of HIV testing, linkage to and retention in HIV care using a community, cluster randomized trial.

DETAILED DESCRIPTION:
Eight of 16 intervention naïve communities in the Agincourt HDSS will be randomized to receive the CM intervention to activate TasP based on the investigators CM conceptual framework. The 16 villages will be randomized based on the "restricted randomization" approach, a stratification method to ensure overall balance between intervention and control communities.

Intervention activities will map onto the investigators six mobilization domains identified in the investigators preliminary work as key components for communities to mobilize for change around HIV prevention. These activities will support communities to: 1) identify a shared concern around testing, linkage and retention in care; 2) enable communities to develop critical consciousness around TasP; 3) facilitate identification and development of structures and networks to disseminate information and activities around TasP; 4) identify and engage community leadership around TasP; 5) take collection action to support TasP; and 6) build community cohesion to address the HIV epidemic and support access to care.

The investigators will evaluate the impact of the intervention using a linked data set including electronic clinic records and the HDSS census data, which will allow us to determine whether people in the intervention communities test at higher proportions than those in control communities, whether individuals who test positive in the intervention communities are more likely to receive CD4 testing and initiate treatment within 3 months than the control communities, and whether those who are eligible and not eligible for treatment are retained in care.

The investigators will implement a representative cross-sectional survey in all 16 villages prior to and following the intervention in order to examine changes in CM domains across villages and the mechanisms through which the intervention affects HIV testing, linkage and retention.

In addition, intervention progress and dosage will be carefully monitored through a tracking system to document all workshops and activities that are carried out in each village.

ELIGIBILITY:
Inclusion Criteria:

* lived in the study area for 12 months
* age 18-49 years
* able to provide informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2338 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Rates of HIV Testing | 3 years follow-up
  Tested /Untested past 12 mos, among HIV-negative or unknown status residents
Rates of linkage to care CD4 within 3 months | 3 years follow-up
  Received CD4 results or had clinical visit within 3 mos of testing HIV positive among recent positives
Rates of retention in care | 3 years follow-up
  No treatment default (no more than a 90-day gap in medication or visit schedule)

SECONDARY OUTCOMES:
Median CD4 of people initiating ART | 3 years follow-up
  Median CD4 at entry into care
Re-engagement in care | 3 years follow-up
  Patients out of care for ≥ 12 months who are re-engaged in care, as evidenced by a clinical visit or CD4 test
Testing Yield | 3 years follow-up
  Number of new diagnoses
First Time Testers | 3 years follow-up
  Number of first time testers (in particular the number of HIV infected undiagnosed)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Pettifor, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- MRC/Wits Rural Public Health and Heath Transitions Research Unit, Agincourt, Mpumalanga, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lippman SA, Pettifor A, Dufour MK, Kabudula CW, Twine R, Peacock D, Mathebula R, Julien A, West R, Neilands TB, Wagner R, Gottert A, Gomez-Olive FX, Rebombo D, Haberland N, Pulerwitz J, Majuba LP, Tollman S, Kahn K. A community mobilisation intervention to improve engagement in HIV testing, linkage to care, and retention in care in South Africa: a cluster-randomised controlled trial. Lancet HIV. 2022 Sep;9(9):e617-e626. doi: 10.1016/S2352-3018(22)00192-8. PMID 36055294
- [Derived] Lippman SA, Pettifor A, Rebombo D, Julien A, Wagner RG, Kang Dufour MS, Kabudula CW, Neilands TB, Twine R, Gottert A, Gomez-Olive FX, Tollman SM, Sanne I, Peacock D, Kahn K. Evaluation of the Tsima community mobilization intervention to improve engagement in HIV testing and care in South Africa: study protocol for a cluster randomized trial. Implement Sci. 2017 Jan 17;12(1):9. doi: 10.1186/s13012-016-0541-0. PMID 28095904